CLINICAL TRIAL: NCT07174531
Title: Multicenter Clinical Trial to Evaluate the Efficacy and Safety of the Renato® Transcatheter Valve-in-Valve System
Brief Title: Renato® Transcatheter Valve-in-Valve System Multicenter Registry Trial (China)
Acronym: VIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Balance Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYL2020A
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Bioprosthesis Failure
Keywords: Valve-in-Valve; Renato; Aortic Valve Replacement; Tricuspid Valve Replacement; Mitral Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prosthesis Failure Valve Replacement (Experimental): Transcatheter valve-in-valve implantation for patients with degenerated aortic/mitral/tricuspid bioprosthetic valves who are at high-risk to redo surgical valve replacement.
  Interventions: Procedure: Transcatheter valve in Valve implantation

INTERVENTIONS:
Procedure: Transcatheter valve in Valve implantation — Transcatheter valve-in-valve implantation for patients with degenerated aortic/mitral/tricuspid bioprosthetic valves who are at high-risk to redo surgical valve replacement.

SUMMARY:
The Renato® transcatheter valve-in-valve system, developed by Balance Medical, is undergoing a multicenter registry trial across China. The study enrolls patients whose previously implanted surgical or transcatheter bioprosthetic valves have deteriorated and who are at high risk for repeat open-heart surgery. A new bioprosthetic valve is delivered via a transcatheter approach and positioned inside the failing valve, restoring valve function .

ELIGIBILITY:
Inclusion Criteria:

1. Pre-existing bioprosthetic valve with clinically significant structural deterioration (≥ moderate stenosis or regurgitation) in the mitral, aortic, or tricuspid position, mandating re-intervention.
2. Estimated high surgical risk (STS predicted risk of mortality ≥ 8 %) or formal contraindication to redo surgical as confirmed by an independent multidisciplinary heart-team review.

Exclusion Criteria:

1. Small true internal diameter of the failing bioprosthesis deemed unsuitable for valve-in-valve therapy by the independent heart-team.
2. Failed mitral bioprosthesis with estimated post-procedural left-ventricular outflow tract obstruction (LVOTO) gradient ≥ 30 mmHg or LVOTO risk classified as "high" by the independent heart-team.
3. Failed tricuspid bioprosthesis with concomitant severe pulmonary hypertension (systolic pulmonary artery pressure > 60 mmHg).
4. Any additional native or prosthetic valve lesion requiring concomitant surgical intervention, as determined by the independent heart-team.
5. More than trivial paravalvular leak around the failing bioprosthesis.
6. Intracardiac thrombus, mass, or vegetation documented by imaging.
7. Myocardial infarction, coronary-stent implantation, cardiac rhythm-device implantation, stroke, or transient ischemic attack within 30 days before screening.
8. Significant coronary artery disease mandating revascularization.
9. Active infective endocarditis within 6 months of screening.
10. Active infection requiring systemic antibiotic therapy at the time of screening.
11. Life expectancy < 12 months for any non-cardiac condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
All-cause death | 12 months.
  Cardiac and non-cardiac mortality will be captured for all enrolled patients.

SECONDARY OUTCOMES:
Safety Parameters | 12 months
  Incidence of major adverse cardiovascular events (MACE), defined as a composite of myocardial infarction, stroke, permanent pacemaker implantation, or rehospitalization due to heart failure,

CONTACTS AND LOCATIONS:
Locations (1):
- Balance Medical, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen J, Yang Y, Song W, Feng D, Yan Y, Wang C, Wei L. Transcatheter tricuspid valve-in-valve implantation for degenerated surgical bioprosthesis. Catheter Cardiovasc Interv. 2023 Feb 1;101(2):442-448. doi: 10.1002/ccd.30554. Epub 2023 Jan 8. PMID 36617381